CLINICAL TRIAL: NCT02426125
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of Ramucirumab Plus Docetaxel Versus Placebo Plus Docetaxel in Patients With Locally Advanced or Unresectable or Metastatic Urothelial Carcinoma Who Progressed on or After Platinum-Based Therapy
Brief Title: A Study of Ramucirumab (LY3009806) Plus Docetaxel in Participants With Urothelial Cancer
Acronym: RANGE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15679; I4T-MC-JVDC (Other: Eli Lilly and Company); 2014-003655-66 (EudraCT Number)
Record Dates: First submitted 2015-04-21; First posted 2015-04-24 (Estimated); Results first posted 2019-03-08 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Urothelial Carcinoma
Keywords: carcinoma of the bladder; carcinoma of the urethra; carcinoma the of ureter; carcinoma of the renal pelvis; transitional cell carcinoma; transitional cell tumor; RANGE; bladder cancer
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Urethral Neoplasms | interventions — Ramucirumab; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ramucirumab + Docetaxel (Experimental): Ramucirumab (10 milligram/kilogram [mg/kg]) intravenously (IV) plus docetaxel (75 milligram/square meter [mg/m²]) IV on day 1 of each 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: Ramucirumab; Drug: Docetaxel
- Placebo + Docetaxel (Placebo Comparator): Placebo IV plus docetaxel (75 mg/m²) IV on day 1 of each 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: Docetaxel; Drug: Placebo

INTERVENTIONS:
Drug: Ramucirumab — Administered IV
  Other Names: LY3009806
  Arms: Ramucirumab + Docetaxel
Drug: Docetaxel — Administered IV
Drug: Placebo — Administered IV
  Arms: Placebo + Docetaxel

SUMMARY:
The main purpose of this study is to evaluate the safety and efficacy of the study drug ramucirumab in combination with docetaxel in participants with urothelial cancer who failed prior platinum-based therapy.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically or cytologically confirmed, locally advanced or unresectable or metastatic urothelial (transitional cell) carcinoma of the bladder, urethra, ureter, or renal pelvis.
* Had disease progression while on a platinum containing regimen in the first-line setting or within 14 months after completing the first-line platinum regimen. Participants who received treatment with one immune checkpoint inhibitor regimen are eligible (for example Programmed death 1 (PD-1), Programmed death-ligand 1 (PDL1), or CTLA4) and may have a longer interval since prior platinum-containing therapy (≤24 months).
* Have a life expectancy of ≥3 months.
* Have received no more than one prior systemic chemotherapy regimen in the relapsed or metastatic setting. Prior treatment with no more than one prior immune checkpoint inhibitor is permitted and will not be considered as a line of systemic chemotherapy.
* Have measurable disease or nonmeasurable but evaluable disease as defined by Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1).
* Have an Eastern Cooperative Oncology Group (ECOG) of 0 or 1.
* Have adequate hematologic function.
* Have adequate coagulation function.
* Have adequate hepatic function.
* The participant does not have:

  * cirrhosis at a level of Child-Pugh B (or worse)
  * cirrhosis (any degree) and a history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis
* Have adequate renal function as defined by creatinine clearance >30 milliliters/minute.
* Have urinary protein ≤1+ on dipstick or routine urinalysis.
* The participant is willing to provide blood, urine, and tissue samples for research purposes.

Exclusion Criteria:

* Have received more than one prior systemic chemotherapy regimen for metastatic disease.
* Have received prior systemic taxane therapy for transitional cell carcinoma (TCC) of the bladder, urethra, ureter, or renal pelvis in any setting (neoadjuvant, adjuvant, metastatic).
* Have received more than one prior antiangiogenic agent (that is, bevacizumab, sorafenib, sunitinib) for TCC of the urothelium.
* Have received radiation therapy within 4 weeks (≤4 weeks) prior to randomization or has not recovered from toxic effects of the treatment that was given >4 weeks prior to randomization.
* Have a history of uncontrolled hereditary or acquired bleeding or thrombotic disorders.
* Have experienced a Grade ≥3 bleeding event within 3 months (≤3 months) prior to randomization.
* Have uncontrolled intercurrent illness, including, but not limited to symptomatic anemia, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, symptomatic or poorly controlled cardiac arrhythmia, psychiatric illness, or any other serious uncontrolled medical disorders.
* Have experienced any arterial or venothrombotic or thromboembolic events, including, but not limited to myocardial infarction, transient ischemic attack, or cerebrovascular accident, within 6 months (≤6 months) prior to randomization.
* Have known untreated brain metastases, uncontrolled spinal cord compression, or leptomeningeal disease.
* Have human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome-related illness.
* Have undergone major surgery within 28 days (≤28 days) prior to randomization or subcutaneous venous access device placement within 7 days (≤7 days) prior to randomization.
* The participant is pregnant prior to randomization or lactating.
* Have a concurrent malignancy or had another malignancy within 5 years (≤5 years) of study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2015-07-13 (Actual); Primary Completion 2017-04-21 (Actual); Study Completion 2022-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (139):
- United States (33):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - St. Jude Medical Center, Fullerton, California
  - UCLA Medical Center, Los Angeles, California
  - USC Norris Cancer Hospital, Los Angeles, California
  - SMO TRIO -Translational Research, Los Angeles, California
  - Cancer Care Associates Medical Group, Redondo Beach, California
  - University of California, Davis - Health Systems, Sacramento, California
  - Central Coast Medical Oncology Corporation, Santa Monica, California
  - University of Colorado, Aurora, Colorado
  - Pharmatech Oncology Inc, Denver, Colorado
  - St Mary's Hospital Regional Cancer Center, Grand Junction, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Southeast Florida Hematology/Oncology, Fort Lauderdale, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Southeastern Regional Medical Center, Newnan, Georgia
  - The Queen's Medical Center, Honolulu, Hawaii
  - Fort Wayne Oncology & Hematology, Fort Wayne, Indiana
  - Alton Ochsner Medical Center, New Orleans, Louisiana
  - University of Maryland- Biological Sciences, Baltimore, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cornell University Medical College, New York, New York
  - SUNY at Stony Brook, Stony Brook, New York
  - Oncology Hematology Care Inc., Cincinnati, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - SMO Sarah Cannon Research Inst., Nashville, Tennessee
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Inova Comprehensive Cancer Care & Research Institute, Fairfax, Virginia
  - University of Washington Medical Center, Seattle, Washington
- Australia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Adelaide
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Footscray
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Randwick
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Subiaco
- Belgium (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leuven
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wilrijk
- Canada (2):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Toronto
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Vancouver
- Denmark (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Herlev
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Odense
- France (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lyon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montpellier
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rennes
- Germany (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Düsseldorf
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Freiburg im Breisgau
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Homburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jena
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tübingen
- Greece (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heraklion
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pátrai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thessaloniki
- Hungary (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miskolc
- Israel (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haifa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kfar Saba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Petah Tikva
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Tel Aviv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tel Litwinsky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ẕerifin
- Italy (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arezzo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bologna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orbassano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Verona
- Japan (17):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bunkyō City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hidaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hirosaki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kashiwa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kita-gun
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kobe
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Matsuyama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morioka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Niigata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sapporo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sendai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suita-shi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tsukuba
- Mexico (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aguascalientes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Culiacán
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., México
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morelia
- Netherlands (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amsterdam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arnhem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Maastricht
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rotterdam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sittard
- Poland (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wieliszew
- Romania (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baia Mare
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Craiova
- Russia (5):
  - Ivanovo regional clinical oncology dispensary, Ivanovo
  - Republic Oncology Dispensary of MoH of Republic Tatarstan, Kazan'
  - Scientific research oncology institute n.a. P. A. Herzen, Moscow
  - Saint-Petersburg city clinical oncology dispensary, Saint Petersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saratov
- South Korea (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daejeon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seongnam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Seongnam-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
- Spain (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Badajoz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
- Taiwan (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaohsiung City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tainan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
- Turkey (Türkiye) (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ankara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Antalya
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edirne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Istanbul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Malatya
- Ukraine (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dnipropetrovsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyiv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lutsk
- United Kingdom (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bebington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Chelsea
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nottingham
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Southampton
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sutton

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] van der Heijden MS, Powles T, Petrylak D, de Wit R, Necchi A, Sternberg CN, Matsubara N, Nishiyama H, Castellano D, Hussain SA, Bamias A, Gakis G, Lee JL, Tagawa ST, Vaishampayan U, Aragon-Ching JB, Eigl BJ, Hozak RR, Rasmussen ER, Xia MS, Rhodes R, Wijayawardana S, Bell-McGuinn KM, Aggarwal A, Drakaki A. Predictive biomarkers for survival benefit with ramucirumab in urothelial cancer in the RANGE trial. Nat Commun. 2022 Apr 6;13(1):1878. doi: 10.1038/s41467-022-29441-y. PMID 35388003
- [Derived] Mitani S, Chen Y, Inoue K, Mori J, Gao L, Long A, Wakabayashi S. Clinical Impact of a Shortened Infusion Duration of Ramucirumab in Japanese Patients -A Model-Based Approach. Gan To Kagaku Ryoho. 2021 Nov;48(11):1381-1387. PMID 34795131
- [Derived] Necchi A, Nishiyama H, Matsubara N, Lee JL, Petrylak DP, de Wit R, Drakaki A, Liepa AM, Mao H, Bell-McGuinn K, Powles T. Health-related quality of life in the randomized phase 3 study of ramucirumab plus docetaxel versus placebo plus docetaxel in platinum-refractory advanced urothelial carcinoma (RANGE). BMC Urol. 2020 Nov 7;20(1):181. doi: 10.1186/s12894-020-00752-w. PMID 33160359
- [Derived] Petrylak DP, de Wit R, Chi KN, Drakaki A, Sternberg CN, Nishiyama H, Castellano D, Hussain SA, Flechon A, Bamias A, Yu EY, van der Heijden MS, Matsubara N, Alekseev B, Necchi A, Geczi L, Ou YC, Coskun HS, Su WP, Bedke J, Gakis G, Percent IJ, Lee JL, Tucci M, Semenov A, Laestadius F, Peer A, Tortora G, Safina S, Garcia Del Muro X, Rodriguez-Vida A, Cicin I, Harputluoglu H, Tagawa ST, Vaishampayan U, Aragon-Ching JB, Hamid O, Liepa AM, Wijayawardana S, Russo F, Walgren RA, Zimmermann AH, Hozak RR, Bell-McGuinn KM, Powles T; RANGE study investigators. Ramucirumab plus docetaxel versus placebo plus docetaxel in patients with locally advanced or metastatic urothelial carcinoma after platinum-based therapy (RANGE): overall survival and updated results of a randomised, double-blind, phase 3 trial. Lancet Oncol. 2020 Jan;21(1):105-120. doi: 10.1016/S1470-2045(19)30668-0. Epub 2019 Nov 18. PMID 31753727
- [Derived] Petrylak DP, de Wit R, Chi KN, Drakaki A, Sternberg CN, Nishiyama H, Castellano D, Hussain S, Flechon A, Bamias A, Yu EY, van der Heijden MS, Matsubara N, Alekseev B, Necchi A, Geczi L, Ou YC, Coskun HS, Su WP, Hegemann M, Percent IJ, Lee JL, Tucci M, Semenov A, Laestadius F, Peer A, Tortora G, Safina S, Del Muro XG, Rodriguez-Vida A, Cicin I, Harputluoglu H, Widau RC, Liepa AM, Walgren RA, Hamid O, Zimmermann AH, Bell-McGuinn KM, Powles T; RANGE study investigators. Ramucirumab plus docetaxel versus placebo plus docetaxel in patients with locally advanced or metastatic urothelial carcinoma after platinum-based therapy (RANGE): a randomised, double-blind, phase 3 trial. Lancet. 2017 Nov 18;390(10109):2266-2277. doi: 10.1016/S0140-6736(17)32365-6. Epub 2017 Sep 12. PMID 28916371
- See also: A Study of Ramucirumab (LY3009806) Plus Docetaxel in Participants With Urothelial Cancer — https://trials.lilly.com/en-US/trial/97404

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers include participants who are confirmed to be alive at study completion.
Period: Overall Study
Arm/Group | Ramucirumab + Docetaxel | Placebo + Docetaxel
Started | 263 | 267
Received at Least One Dose of Study Drug | 258 | 265
Completed | 46 | 39
Not Completed | 217 | 228
Not completed — Lost to Follow-up | 14 | 12
Not completed — Withdrawal by Subject | 13 | 14
Not completed — Death | 185 | 200
Not completed — Randomized, But Never Treated | 5 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Ramucirumab + Docetaxel: Ramucirumab (10 mg/kg) IV plus docetaxel (75 mg/m²) IV on day 1 of each 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Total: Total of all reporting groups
Arm/Group | Ramucirumab + Docetaxel | Placebo + Docetaxel | Total
Number analyzed (Participants) | 263 | 267 | 530
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (9.9) | 64.8 (9.2) | 64.7 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 52 | 102
  Male | 213 | 215 | 428
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 10 | 23
  Not Hispanic or Latino | 208 | 219 | 427
  Unknown or Not Reported | 42 | 38 | 80
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 54 | 61 | 115
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 203 | 204 | 407
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Romania | 5 | 5 | 10
  Hungary | 5 | 8 | 13
  United States | 17 | 18 | 35
  Japan | 24 | 30 | 54
  Ukraine | 5 | 3 | 8
  United Kingdom | 18 | 24 | 42
  Russia | 18 | 12 | 30
  Spain | 22 | 15 | 37
  Greece | 13 | 13 | 26
  Canada | 4 | 5 | 9
  South Korea | 16 | 9 | 25
  Netherlands | 17 | 18 | 35
  Turkey | 11 | 17 | 28
  Belgium | 6 | 1 | 7
  Taiwan | 13 | 18 | 31
  Denmark | 5 | 6 | 11
  Poland | 4 | 4 | 8
  Italy | 23 | 14 | 37
  Mexico | 3 | 1 | 4
  Israel | 7 | 11 | 18
  Australia | 6 | 6 | 12
  France | 16 | 18 | 34
  Germany | 5 | 11 | 16

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS defined as time from first day of therapy to first evidence of disease progression defined by Response Evaluation Criteria in Solid Tumors (RECIST v1.1) or death from any cause. Progressive Disease (PD) is at least 20% increase in sum of diameters of target lesions, with reference being the smallest sum on study and plus absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. If participant does not have complete baseline disease assessment, then PFS time was censored at date of first dose, regardless of whether or not objectively determined disease progression or death has been observed for participant. If participant is not known to have died or have objective progression as of data inclusion cutoff date for analysis, PFS time was censored at last adequate tumor assessment date.
Time Frame: Randomization to Radiological Disease Progression or Death from Any Cause (Up to 18 Months)
Population: The first randomized participants. Censored participants: Ramucirumab + Docetaxel = 58, Placebo + Docetaxel =38.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ramucirumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 216 | 221
Months | 4.07 [2.96 to 4.47] | 2.76 [2.60 to 2.96]
Statistical Analysis 1: Comparison: Ramucirumab + Docetaxel vs Placebo + Docetaxel; Test type: Superiority; p = 0.0118, Log Rank — Stratified; Hazard Ratio (HR) = 0.757, 95% CI 2-sided [0.607 to 0.943] — Stratified

2. Secondary Outcome: Overall Survival (OS)
Description: OS is the time from the date of randomization to the date of death from any cause. For each participant who is not known to have died as of the data inclusion cutoff date for a particular analysis, OS was censored for that analysis at the last known alive date prior to the data inclusion cutoff date.
Time Frame: Randomization to Date of Death from Any Cause (Up to 31.1 Months)
Population: All randomized participants. Censored participants: Ramucirumab + Docetaxel = 78, Placebo + Docetaxel = 67.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Ramucirumab + Docetaxel: Ramucirumab (10 mg/kg) IV plus docetaxel IV on day 1 of each 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
Arm/Group | Ramucirumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 263 | 267
Months | 9.40 [7.89 to 11.43] | 7.85 [7.00 to 9.30]
Statistical Analysis 1: Comparison: Ramucirumab + Docetaxel vs Placebo + Docetaxel; Test type: Superiority; p = 0.2461, Log Rank — Stratified; Hazard Ratio (HR) = 0.887, 95% CI 2-sided [0.724 to 1.086] — Stratified

3. Secondary Outcome: Percentage of Participants With an Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants who achieve a best overall response of complete response (CR) + partial response (PR). ORR = CR + PR. CR is defined as disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 millimeter (mm). Tumor-marker results must have normalized. PR is at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Best overall response is classified based on the overall responses assessed by study investigators according to RECIST v1.1.
Time Frame: Randomization to Disease Progression (Up to 29.7 Months)
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ramucirumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 263 | 267
percentage of participants | 25.9 [20.6 to 31.1] | 13.9 [9.7 to 18.0]

4. Secondary Outcome: Percentage of Participants With Disease Control Rate (DCR)
Description: DCR is the percentage of participants with a best overall response of CR, PR, or Stable Disease (SD) as per Response using RECIST v1.1. Target lesions - CR: Disappearance of all lesions; any pathological lymph nodes must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of lesions vs the baseline sum. Progressive Disease (PD): At least a 20% increase in the sum of diameters of lesions vs the smallest sum on study (the sum must also demonstrate an absolute increase of at least 5 mm); or the appearance of new lesion(s). SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. Non target lesions - CR: Disappearance of all lesions and normalization of tumor marker levels; all lymph nodes must be non-pathological in size. Non-CR/Non-PD: Persistence of lesion(s) and/or maintenance of abnormal tumor marker levels. PD: Unequivocal progression of existing lesions or the appearance of new lesion(s).
Time Frame: Randomization to Disease Progression (Up to 29.7 Months)
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ramucirumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 263 | 267
percentage of participants | 65.4 [59.7 to 71.1] | 55.1 [49.1 to 61.0]

5. Secondary Outcome: Duration of Response (DoR)
Description: Objective response was achieved if they had a best overall response of CR or PR. Target lesions- CR: Disappearance of all lesions; any pathological lymph nodes have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of lesions vs the baseline sum. PD: At least a 20% increase in the sum of diameters of lesions vs the smallest sum on study(the sum must also demonstrate an absolute increase of at least 5 mm); or the appearance of new lesion(s). Non target lesions - CR: Disappearance of all lesions and normalization of tumour marker levels; all lymph nodes must be non-pathological in size. Non-CR/Non-PD: Persistence of lesion(s) and/or maintenance of abnormal tumor marker levels. PD: Unequivocal progression of existing lesions or the appearance of new lesion(s). If a participant was not known to have died or have radiographically documented PD as of the data inclusion cutoff date, DOR was censored at the date of the last adequate tumor assessment.
Time Frame: Date of Complete Response (CR) or Partial Response (PR) to Date of Objective Disease Progression or Death Due to Any Cause (Up to 28.4 Months)
Population: All randomized participants with CR or PR. Participants censored in Ramucirumab + Docetaxel = 12 and in Placebo + Docetaxel = 5.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ramucirumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 68 | 37
Months | 5.32 [3.94 to 6.87] | 4.17 [3.29 to 5.55]
Statistical Analysis 1: Comparison: Ramucirumab + Docetaxel vs Placebo + Docetaxel; Test type: Superiority; p = 0.189, Log Rank; Hazard Ratio (HR) = 0.740, 95% CI 2-sided [0.473 to 1.158]

6. Secondary Outcome: Time to Deterioration in Quality of Life (QoL) on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) - Global Health Status/ QoL Scale
Description: Time to sustained deterioration was defined as time from randomization to first worsening in QoL with no subsequent non-worsened assessment. Worsening in global health status/QoL was defined as a decrease of ≥10 points on a 100-point scale. If a participant did not report worsening, time to sustained deterioration was censored at date of last non-worsened assessment. Scores for global health status/QoL range from 0 to 100 with; higher scores representing better QoL.
Time Frame: Randomization, 30 Days After Treatment Discontinuation (Up to 18 Months)
Population: All randomized participants. Censored participants: Ramucirumab + Docetaxel = 160, Placebo + Docetaxel = 173.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ramucirumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 263 | 267
Months | 6.87 [4.24 to 8.90] | 4.60 [3.52 to 5.55]
Statistical Analysis 1: Comparison: Ramucirumab + Docetaxel vs Placebo + Docetaxel; Global health status/QoL; Test type: Superiority; p = 0.357, Log Rank — Stratified; Hazard Ratio (HR) = 0.879, 95% CI 2-sided [0.663 to 1.167] — Stratified

7. Secondary Outcome: Change From Baseline on the EuroQol 5-Dimension, 5-Level Questionnaire (EQ-5D-5L) Index Score
Description: The EQ-5D-5L is a standardized instrument for use as a measure of self-reported health status. Participants completed the 5-level (no problem, slight problem, moderate problem, severe problem, and inability or extreme problem), 5-dimension (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) questionnaire concerning their current health state. A unique EQ-5D health state is defined by combining 1 level from each of the 5 dimensions. Scores range from 0 (death) to 1 (perfect health), but scores <0 are possible based on the algorithm.
Time Frame: Randomization, 30 Days After Treatment Discontinuation (Up to 18 Months)
Population: All randomized participants with baseline and 30-day follow-up data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ramucirumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 83 | 102
units on a scale | -0.10 (0.26) | -0.19 (0.26)

8. Secondary Outcome: Change From Baseline on the EuroQol 5-Dimension, 5-Level Questionnaire (EQ-5D-5L) Visual Analogue Scale (VAS)
Description: The EQ-5D-5L is a standardized instrument for use as a measure of self-reported health status. A unique EQ-5D health state is defined by combining 1 level from each of the 5 dimensions. Participants indicated their current health status by marking on a VAS ranging from 100 (best imaginable health state) to 0 (worst imaginable health state).
Time Frame: Randomization, 30 Days After Treatment Discontinuation (Up to 18 Months)
Population: All randomized participants with baseline and 30-day follow-up data.
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Groups:
- Placebo + Docetaxel: Placebo IV plus docetaxel (75 mg/m²) IV ion day 1 of each 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
Arm/Group | Ramucirumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 86 | 105
millimeter (mm) | -7.87 (17.95) | -10.91 (16.77)

9. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Ramucirumab
Description: Cmax of Ramucirumab at the end of ramucirumab infusion.
Time Frame: Cycle 1 and Cycle 9, Day 1: Predose, Postdose
Population: All randomized participants who had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (μg/mL)
Arm/Group | Ramucirumab + Docetaxel
Number analyzed (Participants) | 209
microgram/milliliter (μg/mL)
  Cycle 1 | 199 (28)
  Cycle 9: number analyzed (Participants) | 22
  Cycle 9 | 265 (29)

10. Secondary Outcome: PK: Minimum Concentration (Cmin) of Ramucirumab
Description: Cmin of Ramucirumab following administration every 3 weeks.
Time Frame: Day 1 of Cycle 2, 3, 5 and 9 (Predose and Postdose)
Population: All randomized participants who had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Ramucirumab + Docetaxel
Number analyzed (Participants) | 188
μg/mL
  Cycle 2 | 14.9 (64)
  Cycle 3: number analyzed (Participants) | 146
  Cycle 3 | 23.5 (63)
  Cycle 5: number analyzed (Participants) | 94
  Cycle 5 | 32.5 (70)
  Cycle 9: number analyzed (Participants) | 25
  Cycle 9 | 48.9 (56)

11. Secondary Outcome: Number of Participants With Anti-Ramucirumab Antibodies
Description: Number of participants with positive treatment emergent anti-ramucirumab antibodies was summarized by treatment group.
Time Frame: 29.7 Months
Population: All randomized participants who received at least one dose of study drug at baseline and post-baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Ramucirumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 199 | 213
Participants | 3 | 8

ADVERSE EVENTS:
Time Frame: Up to 64.7 Months
Description: All randomized participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Groups:
- Placebo+Docetaxel: Placebo IV plus docetaxel (75 mg/m²) IV on day 1 of each 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
Arm/Group | Ramucirumab + Docetaxel | Placebo+Docetaxel
All-Cause Mortality (participants affected / at risk) | 193/258 | 209/265
Serious Adverse Events (participants affected / at risk) | 111/258 | 107/265
Other Adverse Events (participants affected / at risk) | 241/258 | 251/265
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Ramucirumab + Docetaxel (N=258) | Placebo+Docetaxel (N=265)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 17 (20) | 13 (14)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Neutropenia (Blood and lymphatic system disorders) | 4 (5) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arteriospasm coronary (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 4 (5)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fistula of small intestine (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 2 (2)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2)
Asthenia (General disorders) | 0 (0) | 2 (2)
Chest pain (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 2 (2) | 2 (2)
Fatigue (General disorders) | 5 (5) | 2 (2)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 3 (3) | 9 (10)
Sudden death (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 1 (1)
Device related infection (Infections and infestations) | 3 (3) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 8 (8)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis (Infections and infestations) | 2 (2) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0)
Sepsis (Infections and infestations) | 7 (7) | 5 (5)
Stoma site abscess (Infections and infestations) | 1 (1) | 0 (0)
Toxic shock syndrome (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 10 (11) | 11 (15)
Urosepsis (Infections and infestations) | 2 (2) | 5 (5)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urostomy complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Blood creatinine increased (Investigations) | 1 (1) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (3) | 2 (3)
Platelet count decreased (Investigations) | 2 (2) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basilar artery thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Device connection issue (Product Issues) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 2 (2)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 1 (1)
Haematuria (Renal and urinary disorders) | 4 (4) | 6 (6)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 3 (3) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 2 (2) | 1 (1)
Female genital tract fistula (Reproductive system and breast disorders) | 1/49 (1) | 0/51 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (8)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 2 (2)
Embolism (Vascular disorders) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Venous occlusion (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Ramucirumab + Docetaxel (N=258) | Placebo+Docetaxel (N=265)
Anaemia (Blood and lymphatic system disorders) | 50 (87) | 76 (140)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 9 (9) | 5 (5)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 8 (25) | 5 (9)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 2 (7) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 18 (36) | 14 (14)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (13) | 3 (3)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 2 (3) | 2 (2)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Right atrial enlargement (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 4 (4)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 3 (3) | 2 (2)
Haemophilia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Ear canal stenosis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 3 (4)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (3) | 1 (1)
Dry eye (Eye disorders) | 3 (3) | 2 (2)
Eczema eyelids (Eye disorders) | 1 (1) | 0 (0)
Eye discharge (Eye disorders) | 1 (1) | 0 (0)
Eye disorder (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 2 (4) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 1 (1)
Eyelid function disorder (Eye disorders) | 1 (1) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 24 (28) | 12 (12)
Ocular discomfort (Eye disorders) | 0 (0) | 1 (1)
Photopsia (Eye disorders) | 1 (1) | 0 (0)
Retinal vascular disorder (Eye disorders) | 0 (0) | 1 (2)
Vision blurred (Eye disorders) | 3 (3) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Vitreous detachment (Eye disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 7 (7) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 20 (26) | 17 (22)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 12 (15) | 10 (10)
Abdominal wall disorder (Gastrointestinal disorders) | 0 (0) | 1 (2)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal inflammation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Angular cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 7 (8) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 35 (46) | 45 (58)
Diarrhoea (Gastrointestinal disorders) | 81 (131) | 56 (81)
Dry mouth (Gastrointestinal disorders) | 11 (13) | 5 (5)
Dyschezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 9 (10) | 7 (7)
Dysphagia (Gastrointestinal disorders) | 6 (6) | 2 (2)
Ectopic gastric mucosa (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (8) | 4 (4)
Gingival atrophy (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Glossitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 3 (3) | 2 (2)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 8 (9) | 2 (2)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hyperchlorhydria (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2) | 1 (1)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip blister (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip dry (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 1 (2)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mucous stools (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 71 (102) | 55 (82)
Obstruction gastric (Gastrointestinal disorders) | 1 (5) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Oral disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral hyperaesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Periodontal disease (Gastrointestinal disorders) | 1 (2) | 2 (2)
Proctalgia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (3)
Rectal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal tenesmus (Gastrointestinal disorders) | 2 (2) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 66 (117) | 30 (36)
Toothache (Gastrointestinal disorders) | 1 (1) | 4 (4)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 41 (62) | 40 (56)
Administration site extravasation (General disorders) | 1 (1) | 0 (0)
Administration site rash (General disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 29 (55) | 24 (38)
Catheter site erythema (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 1 (1) | 4 (4)
Chills (General disorders) | 6 (7) | 9 (12)
Extravasation (General disorders) | 0 (0) | 1 (2)
Face oedema (General disorders) | 3 (3) | 1 (1)
Fatigue (General disorders) | 98 (186) | 106 (188)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 2 (2)
Generalised oedema (General disorders) | 1 (2) | 0 (0)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 14 (15) | 7 (7)
Infusion site extravasation (General disorders) | 4 (4) | 0 (0)
Infusion site reaction (General disorders) | 1 (2) | 0 (0)
Injection site extravasation (General disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 5 (12) | 1 (1)
Localised oedema (General disorders) | 1 (2) | 6 (6)
Malaise (General disorders) | 18 (31) | 10 (16)
Moaning (General disorders) | 0 (0) | 1 (1)
Mucosal disorder (General disorders) | 1 (2) | 0 (0)
Mucosal inflammation (General disorders) | 13 (26) | 4 (7)
Nodule (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 4 (4) | 4 (6)
Oedema (General disorders) | 3 (3) | 1 (1)
Oedema peripheral (General disorders) | 38 (52) | 34 (44)
Pain (General disorders) | 10 (14) | 8 (8)
Peripheral swelling (General disorders) | 2 (3) | 0 (0)
Pyrexia (General disorders) | 44 (66) | 42 (63)
Swelling (General disorders) | 2 (2) | 1 (1)
Swelling face (General disorders) | 2 (2) | 1 (1)
Tenderness (General disorders) | 0 (0) | 1 (1)
Thirst decreased (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic pain (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 1 (1)
Allergy to arthropod sting (Immune system disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (2) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (2) | 4 (5)
Seasonal allergy (Immune system disorders) | 1 (1) | 1 (1)
Abscess intestinal (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bacteriuria (Infections and infestations) | 0 (0) | 1 (1)
Breast cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 4 (4) | 3 (3)
Cellulitis (Infections and infestations) | 2 (3) | 2 (2)
Conjunctivitis (Infections and infestations) | 5 (6) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 2 (2) | 1 (1)
Dacryocystitis (Infections and infestations) | 1 (2) | 0 (0)
Device related infection (Infections and infestations) | 2 (2) | 0 (0)
Enterovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 2 (2)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 4 (4) | 2 (2)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes dermatitis (Infections and infestations) | 1 (1) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 1 (2)
Herpes zoster (Infections and infestations) | 2 (2) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Infective glossitis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 1 (1)
Nail bed infection (Infections and infestations) | 1 (3) | 0 (0)
Nail infection (Infections and infestations) | 5 (7) | 1 (1)
Nasopharyngitis (Infections and infestations) | 5 (5) | 3 (3)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (2)
Oral candidiasis (Infections and infestations) | 5 (5) | 3 (3)
Oral fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 2 (3) | 0 (0)
Parotitis (Infections and infestations) | 1 (1) | 0 (0)
Perineal abscess (Infections and infestations) | 0 (0) | 1 (2)
Perineal infection (Infections and infestations) | 1 (2) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (2) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 3 (5)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (2) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 3 (5) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2)
Skin infection (Infections and infestations) | 1 (1) | 1 (1)
Spinal cord infection (Infections and infestations) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 2 (2) | 0 (0)
Tooth infection (Infections and infestations) | 3 (3) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 9 (9)
Urethritis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 31 (38) | 34 (39)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Eschar (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 7 (9) | 6 (6)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nail injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Penis injury (Injury, poisoning and procedural complications) | 0/209 (0) | 1/214 (1)
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stoma site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 9 (9) | 8 (8)
Aspartate aminotransferase increased (Investigations) | 11 (12) | 9 (9)
Blood alkaline phosphatase (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 4 (4) | 11 (14)
Blood bilirubin increased (Investigations) | 2 (6) | 1 (1)
Blood calcium decreased (Investigations) | 0 (0) | 1 (1)
Blood creatine increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 8 (8) | 21 (31)
Blood lactate dehydrogenase increased (Investigations) | 2 (2) | 0 (0)
Blood pressure decreased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 3 (9) | 3 (7)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 2 (2)
Blood uric acid increased (Investigations) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 1 (1) | 0 (0)
Carbon dioxide decreased (Investigations) | 2 (3) | 0 (0)
Clostridium test positive (Investigations) | 1 (1) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 1 (2)
Electrocardiogram st segment depression (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 10 (13)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 5 (15) | 8 (26)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 29 (93) | 29 (71)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 21 (56) | 6 (9)
Platelet count increased (Investigations) | 0 (0) | 1 (1)
Protein total increased (Investigations) | 1 (1) | 0 (0)
Protein urine (Investigations) | 1 (1) | 0 (0)
Protein urine present (Investigations) | 1 (4) | 0 (0)
Prothrombin time prolonged (Investigations) | 1 (1) | 0 (0)
Total lung capacity decreased (Investigations) | 0 (0) | 1 (1)
Troponin t increased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 23 (26) | 21 (28)
Weight increased (Investigations) | 1 (1) | 3 (3)
White blood cell count decreased (Investigations) | 19 (77) | 21 (54)
White blood cell count increased (Investigations) | 0 (0) | 1 (1)
White blood cells urine (Investigations) | 1 (1) | 0 (0)
White blood cells urine positive (Investigations) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 82 (128) | 64 (82)
Dehydration (Metabolism and nutrition disorders) | 8 (8) | 5 (5)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 6 (11) | 12 (15)
Hyperglycaemia (Metabolism and nutrition disorders) | 8 (12) | 13 (15)
Hyperkalaemia (Metabolism and nutrition disorders) | 12 (26) | 7 (12)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 10 (11) | 15 (17)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 17 (25) | 26 (32)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 5 (7)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (4) | 5 (7)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (10) | 10 (11)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 6 (10) | 7 (8)
Vitamin d deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 (39) | 26 (34)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 29 (36) | 21 (26)
Bone pain (Musculoskeletal and connective tissue disorders) | 15 (15) | 17 (19)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (6)
Groin pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 7 (7)
Inguinal mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (4) | 4 (4)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 (6) | 6 (7)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 24 (39) | 23 (30)
Myofascitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (7)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (15) | 16 (22)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pubic pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sacral pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 9 (13)
Ageusia (Nervous system disorders) | 0 (0) | 3 (3)
Amnesia (Nervous system disorders) | 1 (1) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Clonus (Nervous system disorders) | 0 (0) | 1 (2)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (3)
Disturbance in attention (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 7 (8) | 9 (9)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1)
Drooling (Nervous system disorders) | 0 (0) | 1 (1)
Dysaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 28 (41) | 18 (19)
Head titubation (Nervous system disorders) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 19 (27) | 14 (15)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 3 (3)
Hypotonia (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 3 (3) | 1 (1)
Memory impairment (Nervous system disorders) | 2 (2) | 1 (1)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 7 (9) | 13 (16)
Neurotoxicity (Nervous system disorders) | 3 (3) | 2 (2)
Paraesthesia (Nervous system disorders) | 5 (7) | 14 (15)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 18 (23) | 22 (31)
Peroneal nerve palsy (Nervous system disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Taste disorder (Nervous system disorders) | 2 (2) | 1 (1)
Tremor (Nervous system disorders) | 2 (3) | 3 (4)
Device occlusion (Product Issues) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 6 (6) | 8 (10)
Confusional state (Psychiatric disorders) | 1 (1) | 3 (4)
Delirium (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 3 (3) | 4 (4)
Depressive symptom (Psychiatric disorders) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1)
Emotional distress (Psychiatric disorders) | 0 (0) | 1 (1)
Euphoric mood (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 23 (25) | 10 (11)
Irritability (Psychiatric disorders) | 2 (2) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Sleep talking (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 5 (5) | 0 (0)
Anuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder pain (Renal and urinary disorders) | 1 (1) | 1 (1)
Chromaturia (Renal and urinary disorders) | 1 (1) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystitis interstitial (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 3 (3) | 4 (4)
Haematuria (Renal and urinary disorders) | 30 (48) | 19 (20)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydroureter (Renal and urinary disorders) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 2 (2) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 3 (3) | 4 (4)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 33 (60) | 16 (28)
Renal failure (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal impairment (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal pain (Renal and urinary disorders) | 1 (1) | 1 (1)
Urethral haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary fistula (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 6 (6)
Urinary retention (Renal and urinary disorders) | 1 (1) | 5 (6)
Urinary tract obstruction (Renal and urinary disorders) | 2 (2) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 2 (2)
Urine odour abnormal (Renal and urinary disorders) | 1 (1) | 2 (2)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Female genital tract fistula (Reproductive system and breast disorders) | 1/49 (1) | 0/51 (0)
Genital haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (3)
Genital ulceration (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 1/209 (1) | 1/214 (1)
Intermenstrual bleeding (Reproductive system and breast disorders) | 1/49 (2) | 0/51 (0)
Oedema genital (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Pelvic discomfort (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Pelvic organ prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 5 (5) | 4 (4)
Penile pain (Reproductive system and breast disorders) | 0/209 (0) | 1/214 (1)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Perineal ulceration (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Scrotal oedema (Reproductive system and breast disorders) | 3/209 (3) | 1/214 (1)
Scrotal pain (Reproductive system and breast disorders) | 3/209 (3) | 0/214 (0)
Scrotal swelling (Reproductive system and breast disorders) | 0/209 (0) | 1/214 (1)
Testicular oedema (Reproductive system and breast disorders) | 0/209 (0) | 1/214 (1)
Testicular pain (Reproductive system and breast disorders) | 1/209 (1) | 1/214 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1/49 (1) | 1/51 (1)
Vulval haemorrhage (Reproductive system and breast disorders) | 1/49 (1) | 0/51 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1/49 (1) | 0/51 (0)
Aphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (30) | 26 (29)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 32 (50) | 34 (40)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 39 (56) | 14 (16)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 14 (21) | 8 (8)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 5 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 6 (6)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tracheal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 66 (79) | 94 (115)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 11 (12) | 6 (6)
Eczema (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0)
Epidermolysis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 6 (7) | 3 (3)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Nail bed disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 7 (7) | 15 (15)
Nail disorder (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 6 (7) | 3 (3)
Nail toxicity (Skin and subcutaneous tissue disorders) | 2 (4) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Onychalgia (Skin and subcutaneous tissue disorders) | 1 (5) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 5 (7) | 2 (3)
Onychomadesis (Skin and subcutaneous tissue disorders) | 8 (10) | 5 (5)
Pain of skin (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 19 (28) | 6 (15)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (11) | 12 (17)
Rash (Skin and subcutaneous tissue disorders) | 11 (14) | 15 (18)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4)
Xeroderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Catheter placement (Surgical and medical procedures) | 1 (1) | 0 (0)
Central venous catheterisation (Surgical and medical procedures) | 1 (1) | 1 (1)
Endodontic procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
Nail operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Paracentesis (Surgical and medical procedures) | 1 (1) | 0 (0)
Skin lesion removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1)
Cyanosis (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 4 (4)
Embolism (Vascular disorders) | 0 (0) | 2 (2)
Flushing (Vascular disorders) | 4 (5) | 2 (2)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 2 (2) | 2 (2)
Hyperaemia (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 34 (66) | 15 (22)
Hypotension (Vascular disorders) | 7 (10) | 8 (8)
Lymphocele (Vascular disorders) | 1 (1) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1) | 2 (2)
Pallor (Vascular disorders) | 1 (1) | 0 (0)
Pelvic venous thrombosis (Vascular disorders) | 0 (0) | 1 (2)
Phlebitis (Vascular disorders) | 2 (3) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0)
Vasculitis (Vascular disorders) | 1 (6) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Venous occlusion (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2015-01-14): https://cdn.clinicaltrials.gov/large-docs/25/NCT02426125/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-13): https://cdn.clinicaltrials.gov/large-docs/25/NCT02426125/SAP_002.pdf